CLINICAL TRIAL: NCT06456697
Title: Pipeline Embolization Device for the Treatment of Intracranial Aneurysms-A Real World Study on the Long Term Safety and Efficacy(POWER)
Brief Title: Pipeline Embolization Device for the Treatment of Intracranial Aneurysms on the Long Term Safety and Efficacy
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Beijing Tiantan Hospital (Other); Qilu Hospital of Shandong University (Other); Nanfang Hospital, Southern Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: KS2023004
Record Dates: First submitted 2024-05-26; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Treatment
Keywords: intracranial aneurysm; Pipeline
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since its launch in China in 2014, Pipeline Embolization Device (PED) has been widely used in the treatment of intracranial aneurysms. It is necessary to collect data on the long-term safety and efficacy of the Pipeline Embolization Device (PED) in the treatment of intracranial aneurysms, analyze its long-term effectiveness, and provide guidance for clinical practice.

DETAILED DESCRIPTION:
Intracranial aneurysm treatment mainly includes craniotomy clipping and endovascular therapy. In recent years, endovascular treatment techniques have rapidly advanced, especially with the introduction of flow-diverting devices, which have elevated the treatment of intracranial aneurysms to a new level. Different from previous treatment concepts, flow-diverting devices innovate by reconstructing the blood flow in the feeding artery. This reduces the flow velocity and volume entering the aneurysm sac, promotes thrombosis formation inside the aneurysm sac, and induces endothelial growth at the neck of the aneurysm. This approach aims to achieve the goal of aneurysm treatment.

The Pipeline for uncombable or failed aneurysms study (PUFS) results from North America show that the complete occlusion rates at 180 days, 1 year, 3 years, and 5 years follow-up for treating complex intracranial aneurysms with the Pipeline device were 73.6%, 86.8%, 93.4%, and 95.2%, respectively. The rates of significant complications were 5.6%, 1%, 3.5%, and 0%, respectively. The International Retrospective Study of the Pipeline Embolization Device (IntrePED) is a large-scale real-world research conducted in Europe and the United States. It has an average follow-up duration of 19.3 months (1.6 years) and shows an overall complication rate and mortality rate of 8.4%.The results of the single-center prospective PEDESTRIAN registry study at the 5-year follow-up revealed a complete aneurysm occlusion rate of 96.4% and an overall rate of neurological complications, disabilities, and mortality of 5.8%. Based on the current published research findings, there is currently a lack of a multicenter, large-scale study on the long-term safety and effectiveness of the Pipeline flow diversion device for treating intracranial aneurysms internationally.

In China, the pipeline flow diversion device has been in use since 2014, with thousands of reported cases to date. Among them, a significant number of intracranial aneurysm implant devices have been in place for over 5 years. However, there is limited research data available on these cases in China. The most comprehensive study is the Post-Market Multicenter Retrospective Research on Embolization Device in China (PLUS) study, with an average follow-up time of 8.96 ± 7.5 months. The study demonstrated a complete occlusion rate of 81.4% and a complication rate of 4.4%. However, the study primarily focuses on the short to medium-term safety and efficacy, with a current lack of long-term related research.

Therefore, this study aims to collect real-world data on patients with Pipeline embolization devices implanted in a real-world setting. Through analysis, investigators aim to gather real-world evidence on the long-term safety and effectiveness of the Pipeline embolization device for patients with intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was diagnosed with intracranial aneurysms using digital subtraction angiography (DSA).
2. The pipeline was successfully placed to treat intracranial aneurysms.

Exclusion Criteria:

1. Patients had undergone surgery or interventional treatment before enrollment.
2. During treatment, other types of stents are used in combination.
3. Unable to complete the follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted in 10 centers in the country. According to previous literature, the reported occlusion rate ranges from 81.4% to 95.2% [8-12], and the occlusion rate increases with longer follow-up time. In this study, the occlusion rate was calculated at 90%, with a permissible error control of 3%. With α=0.05, the sample size was calculated to be 385. Anticipating a dropout rate of 20%, the sample size needed is 482 cases.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete aneurysm occlusion in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of flow diverter treated cerebral aneurysms (class I: complete obliteration, class II: residual neck, class III: residual aneurysm). Higher class represent a worse outcome. The percentage of Success aneurysm occlusion in which class 1 or 2 is achieved on the Raymond-Roy occlusion classification Scale at the 5 year follow-up angiographic assessments will be evaluated.
Rate of parent artery stenosis in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  Severe stenosis is defined as stenosis greater than 50%.
Patient prognosis in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  Assessing patient prognosis using Modified Rankin Scale (mRS) scores. mRS is scored on a scale of 0 to 6, with a higher score indicating a more severe condition.

SECONDARY OUTCOMES:
Device-related neurologic adverse event in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  This includes but is not limited to shortening, narrowing, and displacement of blood flow devices.
Occurrence of major stroke or neurovascular death in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  This includes but is not limited to ruptured aneurysm, intracerebral hemorrhage on the same side, ischemic stroke, symptomatic stenosis of the feeding artery, and other permanent neurological impairments.
Brain Vascular Accident Leading to Death in 5 years | assessed at 5 years (plus or minus 6 months)after procedure
  Due to other vascular accidents, death occurred.

CONTACTS AND LOCATIONS:
Overall Officials: peng zhang, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China